CLINICAL TRIAL: NCT02540850
Title: Screening of Colorectal Cancer Using Improved SEPT9 (Septin 9) Gene Methylation Assay in Chinese Population
Brief Title: CRC Screening Using mSEPT9 (Methylated Septin 9) in Chinese Population
Acronym: RESEPT
Status: Completed | Type: Observational
Sponsor: BioChain (Beijing) Science and Technology, Inc. (Industry)
Collaborators: Peking Union Medical College Hospital (Other); General Hospital of Beijing PLA Military Region (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RESEPT
Record Dates: First submitted 2015-08-12; First posted 2015-09-04 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Cancer; Adenomatous Polyp of Colon; Polyps; Other Disease/Injury; Other Cancers
Keywords: septin 9; SEPT9; colorectal cancer; CRC; screening; methylation; adenoma; polyps; FIT; FOBT; colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Disease; Wounds and Injuries; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CRC group: stage 0-IV CRC subjects
- precancerous disease group: subjects with adenoma or polyps
- other disease group: subjects with other bowel diseases, other cancers, and subjects with no evidence of disease

SUMMARY:
The purpose of this study is to evaluate the performance of the SEPT9 gene methylation assay in Colorectal cancer (CRC) high-risk population in Chinese hospitals using the opportunistic screening method. The trial plans to evaluate a Chinese domestic SEPT9 assay kit produced by BioChain (Beijing) Science and Technology Corporation, who is a close partner of Epigenomics AG, the producer for Epi proColon 2.0 CE.

DETAILED DESCRIPTION:
1. Background

   Colorectal cancer (CRC) is the third most common malignancy of the gastrointestinal system. Regular screening, early detection and early treatment of colorectal cancer can achieve better prevention and even cure. Currently, 60%-70% of CRC patients are not diagnosed until late stages and only 11.8% of cases are detected at early stage. It is therefore urgent to reduce the CRC mortality by improving the early screening rate. In China,fecal occult blood test (FOBT) and colonoscopy are available presently for early CRC screening. FOBT is widely used due to its low cost and non-invasiveness, however, its false positive rate is relatively high due to many interfering factors. The more advance FOBT, fecal immunochemical test (FIT), has greatly improved the test specificity compared with the traditional chemical method and its compliance is high, but is still subject to the influence of other intestinal diseases, leading to low positive predictive value. In contrast, the compliance for colonoscopy is low due to its invasiveness, cost and risk of complications.

   In recent years, the plasma-based SEPT9 gene methylation assay has proved to be a promising method for the early detection of CRC. Many clinical studies have demonstrated that the methylated SEPT9 gene is a useful biomarker for early CRC detection.At present, Epigenomics' Epi proColon 2.0 CE is the only commercialized assay of SEPT9 gene methylation globally. This product has obtained the approval from the European Union CE certification, the Chinese FDA and the Argentina FDA. It has completed key clinical data submission to the US FDA, with reasonable expectation of the US FDA approval soon. Services based on the SEPT9 gene methylation assay are also provided in clinical laboratories such as quest, Arup, companion to DX and gamma dynacare with the common medical procedure code (CPT code) 81401. In China, BioChain (Beijing) Science and Technology, Inc, a strong partner of Epigenomics AG, has developed its own SEPT9 gene methylation assay with the agreement of Epigenomics AG.
2. Estimation of sample size

   Based on the equation N=Z2* (P (1-p))/E2 for known positivity detection rate, the investigators calculated the number of samples needed for the trial, in which N represents the sample size, Z is a statistical parameter (Z=1.96 for 95% confidence interval); E represents the error (5% was chosen in this study), and P represents the probability (putative positive detection rate). The investigators choose 0.75 for P value based on existing literatures on SEPT9 sensitivity. The number of CRC cases is calculated as 288 based on the equation above. The investigators aim to collect complete information for 300 cases due to information incompleteness and tracking loss. etc. Based on the estimation that CRC account for 30% of high-risk outpatients and inpatients in Chinese hospitals, the total number of patients in the trial should be no less than 1000 cases. The investigators aim at recruiting 1200 cases in this trial taking account of 20% loss of follow-up rate.

   The final actual number of cases for this trial was 1031, due to loss of tracking, incomplete test or clinical data, or samples that did not meet the test criteria.
3. Subject grouping

   All patients will not be grouped before blood draw for SEPT9 assay, and blood samples will be obtained for all subjects who met the selection criteria. All the technicians are blinded to the clinical information of subjects. In order to investigate the feasibility of joint detection with SEPT9 assay and other screening tests, carcino-embryonic antigen (CEA) and FIT tests will be performed at the will of participating patients and the judgment of physicians. This part of data will be used in a retrospective analysis after the completion of the trial.

   When all planned tests are finished, all subjects will be divided into three groups based on colonoscopy diagnosis and pathology, the CRC group, the precancerous disease group and other disease group, in which the CRC group consists of patients with stage 0-IV CRC, the precancerous disease group includes patients of adenoma and polyps, and other disease group includes patients of other bowel disease, other cancers, and subjects with no evidence of disease.
4. Trial procedure

   Training will be finished before the trial starts including the operation procedure of the assay and the use of kits and instruments. This trial is a randomized, single-blind study. All patients should sign the informed consent before blood draw of 10ml. Samples will be processed and the SEPT9 assay will be performed based on the instructions for users. All subjects will receive colonoscopy and/or pathological examination to confirm the diagnosis, and the results for SEPT9 assay will be decided based on the instructions for users. Statistical analysis will be performed based on the results from both SEPT9 assay and colonoscopy and/or pathological examination.
5. Sample collection and storage

1) sample collection:

1. sample should be collected from outpatients or inpatients and the sample information should be recorded in sample collection forms.
2. sample collection: 10 mL peripheral blood (K2EDTA decoagulant only).
3. in order to ensure the accuracy of the assay, sample collection should be performed strictly based on the above requirements, otherwise it may affect the accuracy of the assay.

2) sample storage and transportation method: Store and transfer the samples based on the instructions for use of the kit

6, SEPT9 assay

SEPT9 gene methylation assay (PCR fluorescence probe method) is composed of two steps. Firstly, the cell-free DNA in plasma is extracted using the plasma processing kit, followed by bisulfite conversion, in which the unmethylated cytosine will be converted while the methylated cytosine will not. Secondly, real-time PCR using bisulfite-converted DNA (bisDNA) as the template will be performed to determine the amplification of template. PCR blocking agent and methylation-specific probes can work together to distinguish between methylated and unmethylated DNA. Beta-actin will be used as the internal control to evaluate the plasma DNA quality and the validity of PCR amplification. Positive and negative controls will be provided in the kit as quality controls and will be run parallel with samples each time.

7,Data analysis and statistics

The data for SEPT9 assay and the data of colonoscopy of all subject will be collected and analyzed, the following parameters will be calculated:

Sensitivity Specificity Consistency positive predictive value (PPV) negative predictive value (NPV)

8,Ethics

The budget plan for the clinical trial will be submitted to the ethic committee of participating hospitals for review before the clinical trial starts. The study will not be initiated unless the approval by the committees. All subjects will sign the informed consent before blood collection, and will be informed the usage of plasma and the test results.

9, Research progress

2014.02-2014.04 Confirmation of clinical trial protocols and training of personnel for sample collection and test

2014.04-2014.08 Submission of clinical trial application to ethics committee for approval in four hospitals

2014.08-2015.04 Start patient recruitment and collection of general information of subjects

2014.10-2015.04 Sample collection and tests

2015.04-2015.07 Collect and track the colonoscopy and/or pathology information

2015.07-2015.09 Data processing, statistics and analysis

2015.10 Close of patient recruitment and finish of the trial

10,Budget

The costs include expenses for recruiting 1200 subjects, equipment rent charges, test material costs, sample processing fee, labor costs, patient compensation costs, travel and conference costs, publication and intellectual property (IP) fees. All expenses will be covered by BioChain, as this trial is initiated and organized by BioChain.

11,Publication and intellectual properties

1. plan to publish 2-3 papers in science citation index (SCI)-indexed journals, 3-4 papers in Chinese domestic core journals.
2. plan to submit one patent

12, Data management

Quality of clinical trial data is the basis for evaluation of results. To ensure the reality and reliability of experiment results, the investigators set up a series of data management principles. The investigators will explain data management principles in this study thoroughly in the following from the composition and responsibility of Data Management Committee and content of data management.

13.Research team and personnel

In order to avoid the possible errors caused by difference in disease incidence and ratio of patients in different hospitals, four hospitals in Beijing will be chosen for patient recruitment in this clinical trial. Since patients in these four hospitals are mainly from northern China, the study population is representative for disease epidemiology in this part of the country. Doctors and technicians from the department of gastrointestinal diseases, endoscopy and general surgery from the four hospitals will participate the trial, they are:

Peking Union Medical College Hospital (Beijing) Beijing Military General Hospital (Beijing) Cancer Hospital Chinese Academy of Medical Sciences (Beijing) Beijing Cancer Hospital (Beijing)

ELIGIBILITY:
Inclusion Criteria:

1. sample information is complete, including sample number, gender, age and clinical diagnosis;
2. CRC group: positive samples refer to samples confirmed to be CRC with colonoscopy and/or pathological examination;
3. precancerous disease group: all samples confirmed to be adenoma and polyps by colonoscopy and/or pathological examination
4. other disease group: samples confirmed to be other GI diseases, other cancers or no evidence of diseases by colonoscopy and/or pathological examination

Exclusion Criteria:

1. the patient information is not complete;
2. the sample information is not complete;
3. history of colorectal cancer surgery or other cancer history, or any chemotherapy;
4. women in pregnancy;
5. samples not comply with any of the above selection criteria

Ages: 17 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All eligible inpatients, outpatients, and subjects from health examination centers.
Sampling Method: Probability Sample
Enrollment: 1031 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: XIAOLIANG HAN, Ph.D., Study Director — BioChain (Beijing) Science and Technology, Inc.
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - General Hospital of Beijing PLA Military Region, Beijing
  - Peking Union Medical College Hospital, Beijing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Started | 360 | 396 | 444
Completed | 291 | 330 | 410
Not Completed | 69 | 66 | 34
Not completed — Lost to Follow-up | 69 | 66 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group | Total
Number analyzed (Participants) | 291 | 330 | 410 | 1031
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 188 | 265 | 390 | 843
  >=65 years | 103 | 65 | 19 | 187
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [25 to 88] | 54.7 [24 to 85] | 48.4 [17 to 82] | 53.5 [17 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 144 | 234 | 486
  Male | 183 | 186 | 176 | 545
Region of Enrollment [Number; unit: participants]
  China | 291 | 330 | 410 | 1031

OUTCOME MEASURES:

1. Primary Outcome: Ct Value (Ct Values From PCR Reaction)
Description: the number of PCR cycles where the amplification signal starts to be observed
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Ct
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
Ct | 38.4 [37.8 to 38.9] | 44.3 [44.1 to 44.5] | 44.6 [44.4 to 44.7]

2. Secondary Outcome: Sensitivity (Sensitivity of mSEPT9 Assay in Detecting Colorectal Cancer)
Description: the ratio of positive cases in all CRC cases
Time Frame: 1 year
Measure: Number; unit: Percentage of positives in disease group
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
Percentage of positives in disease group | 76.6 | 8.2 | 0

3. Secondary Outcome: Specificity (Specificity of mSEPT9 Assay in Non-CRC Diseases and NED (no Evidence of Diseases))
Description: the ratio of negative cases in all non-CRC or NED cases
Time Frame: 1 year
Measure: Number; unit: percentage of true negs in non-CRC group
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
percentage of true negs in non-CRC group | 0 | 0 | 95.9

4. Secondary Outcome: PPV (the Positive Predictive Value of mSEPT9 Assay in the Population)
Description: the ratio of true positive in all positive cases
Time Frame: 1 year
Measure: Number; unit: percentage of true pos in all pos cases
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
percentage of true pos in all pos cases | 83.8 | 0 | 0

5. Secondary Outcome: NPV (the Negative Predictive Value of mSEPT9 Assay in the Population)
Description: the ratio of true negative in all negative cases
Time Frame: 1 year
Measure: Number; unit: percentage of true negs in all neg cases
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
percentage of true negs in all neg cases | 0 | 0 | 91.1

6. Secondary Outcome: Positivity Rate (The Ratio of Positive mSEPT9 Results in the Population)
Description: the ratio of positive cases in all cases
Time Frame: 1 year
Measure: Number; unit: percentage of positives in each group
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
percentage of positives in each group | 76.6 | 8.2 | 3.9

7. Secondary Outcome: Consistency (the Overall Ratio of True Positive and True Negative)
Description: The overall consistency ratio of true positive and true negative, i.e. (true positive+true negative)/total number of cases
Time Frame: 1 year
Measure: Number; unit: percentage of true pos&negs in all cases
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Number analyzed (Participants) | 291 | 330 | 410
percentage of true pos&negs in all cases | 89.2 | 89.2 | 89.2

ADVERSE EVENTS:
Arm/Group | CRC Group | Precancerous Disease Group | Other Disease Group
Serious Adverse Events (participants affected / at risk) | 0/291 | 0/330 | 0/410
Other Adverse Events (participants affected / at risk) | 0/291 | 0/330 | 0/410

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement between the sponsor and the clinical hospitals was signed and will be valid if no parties propose to change the agreement, the detailed trial data will not be made public until the trial data is published by the sponsor and/or the hospitals.